CLINICAL TRIAL: NCT05551975
Title: Growth and Tolerance of Preterm Infants Fed an Experimental Human Milk Fortifier
Brief Title: Preterm Infants Fed a Human Milk Fortifier
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AL46
Record Dates: First submitted 2022-09-01; First posted 2022-09-23 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Growth
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Product (Active Comparator): Control Human Milk Fortifier added to human milk feedings
  Interventions: Other: Control Product
- Product 1 (Experimental): Study Human Milk Fortifier added to human milk feedings
  Interventions: Other: Experimental Product 1
- Product 2 (Experimental): Study Human Milk Fortifier added to human milk feedings
  Interventions: Other: Experimental Product 2

INTERVENTIONS:
Other: Control Product — Fed from Study Day 1
  Arms: Control Product
Other: Experimental Product 1 — Fed from Study Day 1
  Arms: Product 1
Other: Experimental Product 2 — Fed from Study Day 1
  Arms: Product 2

SUMMARY:
This is a double-blind, randomized, multi-center, controlled, parallel study to evaluate the growth and tolerance of preterm infants fed human milk fortifier (HMF).

ELIGIBILITY:
Inclusion Criteria:

* Birth weight between 700 g-1500 g.
* ≤ 32 weeks and 0 days GA at birth.
* Participant has been classified as appropriate for GA (AGA).
* Enteral feeding of human milk must be initiated by 21 days of life (birth date is day of life 0)
* Mother agrees to provide human milk as the exclusive feeding during the study period; use of donor milk is permitted if fortified with study fortifier and use of mother's own milk (when available) is prioritized.
* Parent(s) agrees to allow infant to receive both human milk and study HMF.
* Singleton or twin births only.
* Infant's parent(s) or a LAR has voluntarily signed and dated an ICF, approved by an IRB/IEC and provided HIPAA (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* Enteral feeding of preterm infant formula or HMF for > 7 days.
* Expected to be transferred to another facility within 30 days of randomization.
* Serious congenital abnormalities or underlying disease that may affect growth and development.
* 5-minute APGAR ≤ 4.
* Receiving systemic steroids at time of randomization.
* Receiving probiotics at time of randomization.
* Grade Ill or IV PVH/IVH.
* Dependent on invasive ventilation at time of randomization.
* Maternal incapacity.
* Mother or infant is currently receiving treatment consistent with HIV therapy.
* Documentation of maternal use of alcohol or marijuana during pregnancy that in the opinion of the physician is considered abuse.
* Positive toxicology report for cocaine, opiates, or methamphetamine in mother or infant.
* Infant has a history of major surgery (intra-thoracic or intra-abdominal procedures or other surgery requiring general anesthesia).
* Asphyxia defined as progressive hypoxemia and hypercapnia with significant metabolic acidemia characterized by APGAR score <3 at 10 minutes, seizures within the first 12 hours of life, or a cord blood gas < 7.0 and seizures and/or severe tonic abnormalities in the first 12 hours of life.
* Confirmed NEC (Bell's Stage II or III).
* Confirmed current sepsis.
* Infant has any other condition that, in the opinion of the investigator, precludes participation in the study.
* Participation in another study that has not been approved as a concomitant study by AN.
* Participant has an allergy or intolerance to any ingredient in study fortifier.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Weight | Study Day 1 to Study Day 29 or Hospital Discharge if first
  Weight gain per day

SECONDARY OUTCOMES:
Length | Study Day 1 to Study Day 15 and Study Day 29
  Length gains per week
Length | Study Day 1, 8, 15, 22, 29 and Hospital Discharge
  Attained length in cm
Head Circumference | Study Day 1 to Study Day 15 and Study Day 29
  Head circumference gains per week
Head Circumference (HC) | Study Day 1, 8, 15, 22, 29 and Hospital Discharge
  Attained HC in cm
Weight | Study Day 1, 8, 15, 22, 29 and Hospital Discharge
  Attained weight in grams
Weight | Study Day 1 to Study Day 15
  Weight gain per day
Stool Characteristics | Study Day 1 to Study Day 29
  Percent bloody, black, watery, or hard stools
Feeding Intolerance | Study Day 1 to Study Day 29
  Percent periods NPO, feedings withheld due to gastrointestinal intolerance
Full Enteral Feeds | Study Day 1 to Study Day 29
  Days to achieve full enteral feeds

OTHER OUTCOMES:
Blood Chemistries | Study Day 1 to Study Day 29
  Electrolytes, minerals, BUN, alkaline phosphatase
Medications | Study Day 1 to Study Day 29
  Medication usage including frequency and reason for use
Length of Stay | From birth until Discharge, typically 60 days
  Number of days in hospital
Stool Sample | Study Day 1 to Study Day 29
  Characterization of microbiota, immunity
Blood Sample for Immunity/Inflammation | Study Day 1 to Study Day 29
  Cytokines
Adverse Events | Study Day 1 until Discharge, typically 60 days
  Number of participants with adverse events (AEs) and concurrent expected events

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Reverri, PhD, MS, RD, Study Chair — Abbott Nutrition
Locations (14):
- United States (14):
  - Banner - University Medical Center, Phoenix, Arizona
  - UAMS Medical Center, Little Rock, Arkansas
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - South Miami Hospital, Miami, Florida
  - AdventHealth, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Tufts Medical Center, Boston, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - University of New Mexico Children's Hospital, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Woman's Hospital of Texas, Houston, Texas
  - St. Luke's Baptist Hospital, San Antonio, Texas
  - WVU Medicine Children's Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No